CLINICAL TRIAL: NCT06871163
Title: EFFICACY OF INSPIRATORY MUSCLE TRAINING ASSOCIATED WITH MANUAL TECHNIQUES FOR THE LOWER ESOPHAGEAL SPHINCTER AND DIAPHRAGMATIC RELEASE IN INDIVIDUALS WITH GASTROESOPHAGEAL REFLUX DISEASE: A RANDOMIZED CLINICAL TRIAL
Brief Title: EFFICACY OF INSPIRATORY MUSCLE TRAINING ASSOCIATED WITH MANUAL TECHNIQUES IN INDIVIDUALS WITH GERD
Acronym: GERD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, HELENA MEDEIROS ROCHA, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRGE_TMI_2025
Record Dates: First submitted 2025-02-27; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: inspiratory muscle training (IMT); diaphragmatic release; manual techniques for the lower esophageal sphincter
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group IMT (Experimental): inspiratory muscle training (IMT)
  Interventions: Procedure: inspiratory muscle training
- group IMT +TM (Experimental): inspiratory muscle training (IMT) combined with manual techniques for the lower esophageal sphincter (MTLES) and diaphragmatic release (DRT)
  Interventions: Procedure: inspiratory muscle training (IMT) combined with manual techniques for the lower esophageal sphincter (MTLES) and diaphragmatic release (DRT)
- group placebo (Placebo Comparator): a simulated treatment protocol
  Interventions: Procedure: Controle

INTERVENTIONS:
Procedure: inspiratory muscle training — Volunteers allocated to the Sham group will receive proton pump inhibitor medication at a standard dose of 20 mg Participants will perform home-based IMT with a moderate load set at 50% of maximal inspiratory pressure (PImáx), adjusted weekly during in-person sessions at LACAP-UFPE. Training will use the Powerbreathe® Classic Light device, provided to participants for the study duration. The protocol includes three cycles of 10 explosive respiratory incursions, with one-minute rest intervals, performed twice daily for eight weeks. Participants will record perceived exertion (Borg scale) and any occurrences in a training log.
  Arms: group IMT
Procedure: inspiratory muscle training (IMT) combined with manual techniques for the lower esophageal sphincter (MTLES) and diaphragmatic release (DRT) — Volunteers allocated to the group will receive proton pump inhibitor medication at a standard dose of 20 mg.
  The IMT protocol will be the same as in Group 1. Intervention: IMT Combined with Manual Techniques (MTLES & DRT) The IMT protocol follows Group 1. DRT (Rocha et al., 2015) involves manual traction during inspiration and deepened contact during expiration, applied in two sets of ten deep breaths. MTLES (Eguaras et al., 2019) is performed with the patient seated, applying epigastric pressure to access the lower esophageal sphincter through coordinated flexion-inspiration and extension-expiration for 5 minutes.
  Arms: group IMT +TM
Procedure: Controle — Volunteers allocated to the Sham group will receive proton pump inhibitor medication at a standard dose of 20 mg, as prescribed for other participants. They will undergo a simulated treatment protocol, including inspiratory muscle training (IMT) without load to mimic device use and manual techniques where the therapist places hands on the intervention area without performing actual manipulation.
  Arms: group placebo

SUMMARY:
The objective of this clinical trial is to investigate the efficacy of inspiratory muscle training (IMT) combined with manual techniques for the lower esophageal sphincter (MTLES) and diaphragmatic release (DRT) in patients with Gastroesophageal Reflux Disease (GERD). The main questions it aims to answer are:

1. If the combination of IMT, DRT, and MTLES can improve GERD symptoms and patients' quality of life.
2. If the home-based IMT protocol, with weekly adjustments, and the manual techniques applied twice a week can have a positive impact on various clinical measures, such as pressure at the lower esophageal sphincter, reflux episodes, and quality of life.

The researchers will compare three groups: Group 1 (IMT), Group 2 (IMT + DRT + MTLES), and Group 3 (control, sham), to see if the group receiving IMT combined with DRT and MTLES shows greater improvements compared to the control group.

Participants will perform inspiratory muscle training at home, following a protocol adjusted weekly, and will receive manual techniques twice a week.

DETAILED DESCRIPTION:
The IMT protocol will be performed at home with a load set at 50% of maximal inspiratory pressure (MIP) and adjusted weekly, while manual techniques will be applied twice a week at LACAP. Outcomes include mean pressure at the gastroesophageal junction (esophageal manometry), number of reflux episodes and acid exposure time (impedance-pH monitoring), diaphragmatic mobility and thickness (ultrasound), respiratory muscle strength (manovacuometry), heart rate variability (heart rate monitor), and reflux symptoms and quality of life (questionnaires). It is expected that the combination of IMT, DRT, and MTLES will improve GERD symptoms and positively impact patients' quality of life, providing an effective and less invasive alternative compared to conventional interventions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with gastroesophageal reflux disease (GERD)
* using 20 mg of proton pump inhibitors (PPIs).

Exclusion Criteria:

* Individuals with a hiatal hernia >3 cm,
* chronic lung diseases (chronic obstructive pulmonary disease and interstitial lung diseases)
* severe heart diseases,
* history of previous abdominal and/or thoracic surgeries, rib fractures within the past year,
* severe osteoporosis
* BMI >30 kg/m²

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
pressure at the gastroesophageal junction | Pre-intervention and after 8 weeks of intervention.
  esophageal manometry
number of reflux episodes | Pre-intervention and after 8 weeks of intervention.
  impedance-pH monitoring
reflux symptoms | Pre-intervention and after 8 weeks of intervention.
  Gastroesophageal Reflux Disease Symptom Questionnaire
acid exposure time | Pre-intervention and after 8 weeks of intervention.
  impedance-pH monitoring

SECONDARY OUTCOMES:
diaphragmatic mobility and thickness | Pre-intervention, after 4 weeks of intervention, after 8 weeks of intervention and And a follow-up one month after the last intervention.
  ultrasound
respiratory muscle strength | Pre-intervention, after 4 weeks of intervention, after 8 weeks of intervention and And a follow-up one month after the last intervention.
  manovacuometry
heart rate variability | Pre-intervention, after 4 weeks of intervention, after 8 weeks of intervention and And a follow-up one month after the last intervention.
  heart rate monitor
diaphragmatic thickness | Pre-intervention, after 4 weeks of intervention, after 8 weeks of intervention and And a follow-up one month after the last intervention.
  ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil